CLINICAL TRIAL: NCT02884596
Title: Anesthetic Success of Inferior Alveolar Nerve Block for Mandibular Molars With Symptomatic Irreversible Pulpitis in Women Taking Selective Serotonin Reuptake Inhibitors
Brief Title: Success of Inferior Alveolar Nerve Block in Women Taking Selective Serotonin Reuptake Inhibitors
Status: Completed | Type: Observational
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Masoud Saatchi, DDS MSc, Professor of Endodontics, School of Dentistry, Isfahan University of Medical Sciences, Isfahan University of Medical Sciences
Other Study IDs: 394867
Record Dates: First submitted 2016-08-21; First posted 2016-08-31 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Local Anesthesia
Keywords: Inferior alveolar nerve block; irreversible pulpitis; selective serotonin reuptake inhibitor antidepressants
MeSH Terms: interventions — Selective Serotonin Reuptake Inhibitors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: selective serotonin reuptake inhibitor — Taking any type of SSRI medicaments
  Other Names: SSRI

SUMMARY:
To evaluate the success of inferior alveolar nerve block (IANB) for mandibular molars with irreversible pulpitis in women under treatment with selective serotonin reuptake inhibitors (SSRIs).

DETAILED DESCRIPTION:
Seventy patients with a diagnosis of symptomatic irreversible pulpitis in one mandibular molar were assigned to either SSRI users or SSRI non-users groups. SSRIs users were 45 women who take SSRIs referred for endodontic treatment from a psychiatric clinic to the clinic of the endodontic department of Isfahan University of Medical Sciences. SSRIs non-users were 45 women who did not take SSRIs referred for endodontic treatment to the same dental clinic. The protocol of the study was approved by the Ethics Committee of the university (no. 394867). Written informed consent was obtained from all the patients. The level of anxiety of the patients was determined by using the Corah Dental Anxiety Scale. The patients registered their baseline pain severity using a Heft-Parker visual analogue scale (HP-VAS). Two standard IANBs (1.8-mL cartridges) of 2% lidocaine with 1:100,000 epinephrine (Darupakhsh, Tehran, Iran) were administered to each patient. Fifteen minutes after injection, the teeth were isolated. Access cavity preparation was started. The patients was instructed by the same operator to mark his or her pain experienced during the access cavity preparation.

ELIGIBILITY:
Inclusion Criteria:

* vital mandibular molar tooth
* diagnosis of symptomatic irreversible pulpitis

Exclusion Criteria:

* younger than 18 years old
* history of significant medical conditions
* allergies to local anesthetics or sulfites
* pregnancy
* active sites of pathosis in area of injection
* inability to give informed consent

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Seventy adult women patients participated in this study and were assigned to either SSRIs users or SSRIs non-users groups. SSRIs users were 45 women who take SSRIs referred for endodontic treatment from a psychiatric clinic to the clinic of the endodontic department of Isfahan University of Medical Sciences. SSRIs non-users were 45 women who did not take SSRIs referred for endodontic treatment to the same dental clinic.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2015-06; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
the success rate of the IAN block | taking any type of SSRI for at least six weeks prior to the study

CONTACTS AND LOCATIONS:
Overall Officials: Abbasali khademi, Study Chair — Isfahan University of Medical Sciences
Locations (1):
- School of Dentistry, Isfahan University of Medical Sciences, Isfahan, Iran

IPD SHARING:
Plan to Share IPD: No